CLINICAL TRIAL: NCT00005035
Title: A Phase II Study of Oxaliplatin in Patients With Advanced Carcinoma of the Head and Neck
Brief Title: Oxaliplatin in Treating Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067571; OSU-99H0309; NCI-T99-0016
Record Dates: First submitted 2000-04-06; First posted 2004-03-04 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2002-02

CONDITIONS: Head and Neck Cancer
Keywords: metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of oxaliplatin in treating patients who have advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with advanced squamous cell carcinoma of the head and neck when treated with oxaliplatin. II. Characterize the toxicities and pharmacokinetics of this drug in this patient population. III. Determine the duration of response, time to progression, and survival of these patients receiving this drug.

OUTLINE: Patients are stratified according to prior treatment with neoadjuvant chemotherapy (yes vs no). Patients receive oxaliplatin IV over 2 hours weekly for 4 weeks followed by 2 weeks of rest. Treatment continues every 6 weeks in the absence of unacceptable toxicity or disease progression. Patients are followed until toxicity resolves or for no less than 30 days.

PROJECTED ACCRUAL: A total of 34-74 patients will be accrued for this study within 17 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed squamous cell carcinoma of the head and neck Recurrent or metastatic OR Locally advanced and judged incurable by surgery or radiotherapy Bidimensionally measurable disease New and unirradiated lesion within prior radiation field acceptable as measurable disease if at least 3 months since prior radiotherapy No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 OR Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal AST/ALT no greater than 2.5 times upper limit of normal Renal: Creatinine normal OR Creatinine clearance at least 60 mL/min Cardiovascular: No symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No evidence of neuropathy No history of allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with protocol therapy No other concurrent uncontrolled illness (e.g., ongoing or active infection) Not HIV positive AND receiving antiretroviral therapy (HAART)

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy for head and neck cancer No concurrent colony stimulating factors during first course of therapy Chemotherapy: No prior chemotherapy for recurrent or metastatic disease At least 3 months since prior chemotherapy as initial treatment Endocrine therapy: No prior hormonal therapy for head and neck cancer Radiotherapy: See Disease Characteristics At least 3 months since prior radiotherapy as initial treatment Surgery: See Disease Characteristics Prior surgery allowed Other: No other concurrent investigational or commercial agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris A. Rhoades, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (11):
- United States (11):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Saint Joseph's Regional Medical Center, South Bend, Indiana
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina